CLINICAL TRIAL: NCT05394805
Title: A One-year Non-Interventional Registry to Assess Safety and Effectiveness of HUMIRA® (Adalimumab) in Patients With Moderately to Severely Active Crohn's Disease (CD) in China
Brief Title: A Study of Subcutaneous HUMIRA (Adalimumab) Injection to Assess Adverse Events and Change in Disease Activity In Adult Participants With Moderate to Severe Active Crohn's Disease (CD)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-043
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; HUMIRA®; Adalimumab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants treated with Humira (Adalimumab): Participants prescribed Humira (adalimumab) for moderately to severely active crohn's disease (CD) in routine clinical practice.

SUMMARY:
Crohn's disease (CD) is an incurable chronic inflammatory disorder of the gastrointestinal tract. This study will assess how safe and effective Humira (adalimumab) is in treating moderately to severely active CD in China. Adverse events and change in disease activity will be assessed.

Humira (adalimumab) is a drug approved for the treatment of Crohn's disease (CD).All study participants will receive Humira as prescribed by their study doctor in accordance with approved local label. Approximately 252 participants will be enrolled in China.

Participants will receive subcutaneous HUMIRA (adalimumab) injection as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for 1 year.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants meet the diagnosis of moderate to severe Crohn's disease.
* Participants prescribed with Humira, under investigators' sufficient consideration of benefits/ risks per local label.

Exclusion Criteria:

* Participants who have any of the contraindications as per adalimumab (Humira) label in China.
* Participants who are allergic to any component of adalimumab (Humira).
* Participants with active hepatitis B diagnosed.
* Participants with severe active infection, or known history of active or latent tuberculosis (TB), or latent TB infection with inadequate treatment.
* Participants with cancer diagnosed, excluding also those with non-melanoma skin cancer (NMSC) completely treated, per local label.
* Participants with moderate to severe heart failure.
* Participants who are unwilling to participate, or not suitable for participation as judged by the investigator at risk of noncompliance to study procedure.
* Participants who are enrolled to other interventional studies.
* Participants who are prescribed with adalimumab but choose Humira bio-similar in China.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adult participants with moderately to severely active crohn's disease (CD).
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAEs) | Upto week 52
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.

SECONDARY OUTCOMES:
Number of Participants With Serious Adverse Drug Reaction (ADR) | Upto week 52
  Adverse drug reactions were defined as adverese events (AEs) of which a causal relationship with adalimumab could not be ruled out.
Number of Participants With Non-Serious Adverse Drug Reaction (ADR) | Upto week 52
  Adverse drug reactions were defined as adverese events (AEs) of which a causal relationship with adalimumab could not be ruled out.
Number of Participants who Achieved Clinical Remission Harvey-Bradshaw index (HBI) | Upto week 52
  The HBI is a simplified version of the Crohn's Disease Activity Index(CDAI). The HBI consists of 5 items encompassing patient-reported (well-being, symptoms)and objective (presence of abdominal mass or complications) variables. The total HBI score is the sum of the values for each of the five items. Higher HBI scores indicate greater disease activity. Scores < 5 indicate clinical remission, 5 - 7 indicate mild disease, 8 - 16 indicate moderate disease, and 16 indicate severe disease.
Number of Participants who Achieved Clinical Response Harvey-Bradshaw index (HBI) | Upto week 52
  The HBI is a simplified version of the Crohn's Disease Activity Index(CDAI). The HBI consists of 5 items encompassing patient-reported (well-being, symptoms)and objective (presence of abdominal mass or complications) variables. The total HBI score is the sum of the values for each of the five items. Higher HBI scores indicate greater disease activity. A reduction of 3 points and above is considered as relevant to define clinical response harvey-bradshaw index (HBI).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- China (10):
  - Peking University Third Hospital /ID# 242803, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University /ID# 242798, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 243386, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 242799, Guangzhou, Guangdong
  - Nanjing Drum Tower Hospital /ID# 243385, Nanjing, Jiangsu
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 243213, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 242804, Chengdu, Sichuan
  - Zhejiang Provincial Hospital of Chinese Medicine /ID# 243443, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 242802, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine /ID# 242801, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-043#additional-resources-section